CLINICAL TRIAL: NCT01396499
Title: A Phase I Open-label Study to Assess the Safety, Tolerability and Preliminary Efficacy of BKM120, PI3K Kinase Inhibitor, in Patients With Advanced Leukemias
Brief Title: Study to Assess Safety, Tolerability and Preliminary Efficacy of BKM120, PI3K Kinase Inhibitor, With Advanced Leukemias
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0874; NCI-2011-01610 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-07-15; First posted 2011-07-18 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Leukemia
Keywords: Leukemia; Acute leukemias; Relapsed/refractory leukemias; Acute myelogenous leukemia; AML; Acute lymphoblastic leukemia; ALL; BKM120
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BKM120 (Experimental): Oral BKM120 starting dose 80 mg once daily.
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120 — Starting dose 80 mg tablets by mouth daily for a 28 day cycle.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of BKM120 that can be given to patients with relapsed or refractory leukemia. The safety of BKM120 will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

BKM120 is designed to block a protein that is important to the growth and division of cancer cells, which may cause the cells to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of BKM120 based on when you join this study. Up to 2 dose levels of BKM120 will be tested. Up to six (6) participants will be enrolled at each dose level. The first group of participants will receive the lower dose level.

You will take BKM120 tablets by mouth with a large glass of water every day you are on this study. You should take BKM120 about 1 hour after a light breakfast. You should take BKM120 at about the same time each day. You need to fast (not eat or drink anything except water) for 2 hours after you take your BKM120 dose.

You should swallow the BKM120 tablets whole. The tablets must not be chewed, broken, or crushed. If you vomit after taking BKM120, you should not take another tablet that day to make up for that dose. If you forget to take BKM120 one morning, call your doctor and ask for instructions. Do not take BKM120 after 6pm of the same day or take any extra doses to make up for the missed dose.

If your study doctor feels it is needed or if you have side effects, BKM120 may be stopped and then started again at a lower dose or may be stopped completely.

You will be asked to record in a pill diary each dose you take. You will return the pill diary, unused study drug, and pill containers to the clinic staff at the end of each cycle.

Study Visits:

On this study, each study cycle will last 28 days. You will have study visits every other week (Days 1 and 15) during the first 2 cycles of the study, and then once a month after that. The following tests and procedures will be performed at all study visits:

* Your medical history will be recorded
* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and about any side effects you may be having.
* Blood (about 1 tablespoon) will be drawn for routine tests and to check your blood sugar. ° You will need to fast for 8 hours before this blood draw.
* You will complete the questionnaires about your mood.

On Day 28 of Cycle 1 and every 3 months after that, you will have a bone marrow aspirate and/or biopsy to check the status of the disease. You may have additional bone marrow aspirations collected while you are on study if the doctor thinks they are needed.

Every 4 months, you will have a MUGA scan or an ECHO to check the status of the disease.

ECGs and chest x-rays may be performed throughout the study to check your heart and lung function if the doctor thinks they are needed.

Length of Study:

You may continue taking the study drug for as long as 12 cycles if the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-study visit.

End-of-Study Visit:

After you stop taking BKM120, you will have an end-of-study visit. The following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* You will be asked about any drugs you may be currently taking or have taken.
* You will complete the questionnaires about your mood.
* Blood (about 1 tablespoon) and urine will be collected for routine tests. The blood will also be used to check your kidney and liver function and to check your blood sugar. You will need to fast for 8 hours before this blood draw.
* You will have a MUGA scan or an ECHO to check the status of the disease.
* You will have a bone marrow aspirate and/or biopsy to check the status of the disease.

This is an investigational study. BKM120 is not FDA approved or commercially available. It is currently being used for research purposes only.

Up to 16 patients take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old or older
2. Relapsed/refractory leukemias for which no standard therapy options are anticipated to result in a durable remission: Acute myelogenous leukemia (AML) by World Health Organization (WHO) classification or acute lymphoblastic leukemia (ALL) relapsed or refractory to standard chemotherapy; unsuitable for standard chemotherapy or unwilling to undergo standard chemotherapy. Philadelphia chromosome (Ph) positive ALL eligible if failed prior tyrosine-kinase inhibitor therapy. Age =/> 60 years with AML not candidates for or have refused standard chemotherapy, excluding subjects with acute promyelocytic leukemia (APL) or with favorable cytogenetic abnormalities [inv16, t(8;21)].
3. Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2
4. Serum total bilirubin </= 2 x ULN or direct bilirubin </=ULN for patients with total bilirubin levels > 2 x ULN, unless elevation is thought to be due to hepatic infiltration by AML, Gilbert's syndrome, or hemolysis. Aspartate aminotransferase or alanine aminotransferase within normal range (or =/< 3.0 x upper limit of normal (ULN) if due to leukemic involvement); serum creatinine =/< 1.5 x ULN or 24-hour clearance =/> 50 mL/min; serum amylase </= ULN; serum lipase</= ULN.
5. Fasting glucose =/< 120 mg/dL (6.7 mmol/L).
6. Total calcium (corrected for serum albumin) within normal limits (8.8 - 10.5 MG/DL). This is MD Anderson Cancer Center (MDACC) lab standard. Supplements for calcium allowed to meet eligibility criteria.
7. Magnesium >/= the lower limit of normal (1.8 MG/DL). Supplements for magnesium allowed to meet eligibility criteria
8. Potassium within normal limits (3.5 - 5.0 milliequivalent (MEq)/L). Supplements for potassium allowed to meet eligibility criteria
9. international normalized ratio (INR) =/< 2
10. Women of childbearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum or urine pregnancy test within 48 hours prior to the start of study drug
11. Patients should be able to take oral medications.

Exclusion Criteria:

1. Patients who have received myelosuppressive chemotherapy </= to 4 weeks prior to starting study drug (with the exception of Hydroxyurea which will be allowed during Course 1 of treatment).
2. Patients who have received targeted anticancer therapy ≤ 2 week (for non myelosuppressive therapy) prior to starting study drug.
3. central nervous system (CNS) disease
4. Patient has active cardiac disease including any of the following: Left ventricular ejection fraction (LVEF) < 50% as determined by Multiple Grated acquisition (MUGA) scan or echocardiogram (ECHO), corrected QT interval (QTc) > 480 msec on screening ECG (using the QTcF formula), Angina pectoris that requires the use of anti-anginal medication, Ventricular arrhythmias except for benign premature ventricular contractions, Supraventricular and nodal arrythmias requiring a pacemaker or not controlled with medication, Conduction abnormality requiring a pacemaker, Valvular disease with document compromise in cardiac function, Symptomatic pericarditis
5. Patient has a history of cardiac dysfunction including any of the following: Myocardial infraction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function Documented congestive heart failure (New York Heart Association functional classification III-IV) Documented cardiomyopathy
6. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., e.g., uncontrolled infection, such as persistent fever despite antibacterial therapy) that could cause unacceptable safety risks or compromise compliance with the protocol. Significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of predicted lung volumes, diffusion capacity of lung for carbon monoxide (DLco), O2 saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates.
7. Patient has poorly controlled diabetes mellitus or steroid-induced diabetes mellitus
8. Patients with acute or chronic liver, renal disease or pancreatitis
9. Patients with diarrhea >/= CTCAE grade 2
10. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection). Patients with unresolved diarrhea will be excluded as previously indicated
11. Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) </= 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
12. Patients with the following mood disorders as judged by the Investigator or a psychiatrist, or as a result of patient's mood assessment questionnaire: a. Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others) b. >/= CTCAE grade 3 anxiety c. Meets the cut-off score of >/= 10 in the Patient Health Questionnaire PHQ-9 or a cut-off of >/= 15 in the General Anxiety Disorder GAD-7 mood scale, respectively, or selects a positive response of "1, 2, or 3" to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9) will be excluded from the study unless overruled by the psychiatric assessment
13. Patients who have received prior treatment with a PI3K inhibitor
14. Patients with a known hypersensitivity to BKM120 or to its excipients
15. Patients who are currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug. Please refer to table 4-7 or a list of prohibited QT prolonging drugs with risk of Torsades de Pointes
16. Patients who are currently treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. If treatment with such an inhibitor is in the best interest of the patient, extreme caution should be taken with its concomitant use. Please refer to Table 4-6 for a list of prohibited inhibitors and inducers of CYP3A (Please note that co-treatment with weak inhibitors of CYP3A is allowed)
17. Patients receiving chronic treatment with steroids or another immunosuppressive agent
18. Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug. Herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Fruits include the CYP3A inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits
19. Patients who have undergone major surgery </= 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
20. Patients who are currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant
21. Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control. Double barrier contraceptives must be used through the trial by both sexes. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Women of child-bearing potential must have a negative serum or urine pregnancy test ≤ 48 hours prior to initiating treatment.
22. Known diagnosis of human immunodeficiency virus (HIV) infection
23. History of another malignancy within 3 years, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix and squamous cell carcinoma in situ of the skin.
24. Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of BKM 120 | 28 days, Cycle 1
  Maximum tolerated dose (MTD) defined as highest dose in which 1/6 or less subjects experience a dose limiting toxicity (DLT) during the first course of treatment.
  Toxicity assessed using the NCI Common Toxicity Criteria for Adverse Events, version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Konopleva, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org